CLINICAL TRIAL: NCT03184454
Title: Combined Cortical and Subcortical Recording and Stimulation as a Circuit-Oriented Treatment for Obsessive-Compulsive Disorder
Brief Title: Combined Cortical/Subcortical Recording and Stimulation as a Circuit-Oriented Treatment for Obsessive-Compulsive Disorder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Cristina Cusin, MD, Associate Professor in Psychiatry, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000456
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obsessive Compulsive Disorder
Keywords: OCD; deep brain stimulation; treatment-resistant OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Cortical and subcortical electrodes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic Percept Deep Brain Stimulation (Experimental): Single open label arm.
  Patients with severe, treatment-refractory obsessive-compulsive disorder (OCD) will receive stimulation in two separate, but related, brain regions, the dorsolateral prefrontal cortex (dlPFC) and the ventral anterior limb of the internal capsule and adjacent ventral striatum (VC/VS) with a novel Medtronic Percept deep brain stimulation (DBS) system.
  Interventions: Device: Medtronic Percept Deep Brain Stimulation

INTERVENTIONS:
Device: Medtronic Percept Deep Brain Stimulation — Deep Brain stimulation involves bilateral stereotactic placement of stimulating "leads" into specific brain structures. Leads are attached to permanent subcutaneous wires and battery-powered implantable neurostimulators (INSs). Noninvasive INS programming can achieve a balance between maximal benefit (reduction in disabling OCD symptoms), while minimizing adverse effects (eg sensorimotor effects such as dysarthria or paresthesias; as well as behavioral side effects, e.g., hypomania, insomnia, or increased anxiety).

SUMMARY:
This study involves the use of the Medtronic PC+S deep brain stimulation for the treatment of intractable OCD.

DETAILED DESCRIPTION:
The goal of this proposal is to provide therapy to patients with severe, treatment-refractory obsessive-compulsive disorder (OCD) by stimulating in two separate, but related, brain regions, the dorsolateral prefrontal cortex (dlPFC) and the ventral anterior limb of the internal capsule and adjacent ventral striatum (VC/VS) with a novel Medtronic PC+S deep brain stimulation (DBS) system. While providing this DBS therapy, use of this new, recording-capable device will allow collection of data about brain activity in these two regions. This data will enable researchers to further elucidate the exact mechanisms of DBS therapy, as well as the neuropathophyisiology of OCD. This study aims to 1) gather evidence for corticostriatal changes in OCD in response to acute and chronic VC/VS DBS treatment and 2) specifically disrupt or enhance synchrony in the cortico-striato-thalamo-cortical (CSTC) circuit.

Deep Brain stimulation involves bilateral stereotactic placement of stimulating "leads" into specific brain structures. Leads are attached to permanent subcutaneous wires and battery-powered implantable neurostimulators (INSs). Noninvasive INS programming can achieve a balance between maximal benefit (reduction in disabling OCD symptoms), while minimizing adverse effects (eg sensorimotor effects such as dysarthria or paresthesias; as well as behavioral side effects, e.g., hypomania, insomnia, or increased anxiety). HDE approval was granted in February 2009, and IDE approval was granted in February 2016. Multiple hospitals around the country have established HDE protocols to implant patients with intractable OCD who have failed conventional therapies, and some hospitals, like us, have obtained Investigational Device Exemption (IDE) approval to conduct pilot clinical trials. The existing model of DBS for OCD only addresses one aspect of the brain circuit implicated in the CSTC circuit, the VC/VS target. Therapy with this device, under this protocol, will also be able to provide stimulation to the cortical part of this circuit. Single-site VC/VS DBS may not adequately target the putative circuit. If OCD symptoms do arise from CSTC loop dysfunction, this implies that the problem is one of improper information flow between connected brain areas. Thus, modifying circuit activity may require coordinated intervention at multiple points to effectively synchronize or de-synchronize the full loop. Stimulation that specifically interrupts reverberant activity between prefrontal cortex and striatum will be superior to VC/VS DBS alone at relieving symptoms of OCD. We will test this by simultaneously implanting stimulating/recording electrodes at both VC/VS and a dorsolateral prefrontal cortex (dlPFC) target bilaterally.

ELIGIBILITY:
Inclusion Criteria:

1. OCD, diagnosed by Structured Clinical Interview for DSM-5 (SCID-5), judged of disabling severity with a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 28.
2. Persistence of severe symptoms and impairment for five or more years despite: i. at least three adequate (≥3 months at the maximum tolerated dose) serotonin transporter inhibitor trials (may use any serotonin or serotonin-norepinephrine inhibitors, but must include a trial of clomipramine) alone or in combination with ii. adequate behavior therapy (≥20 sessions of expert exposure and response prevention; At least 20 sessions of behavioral therapy must be attempted), and iii. augmentation of one of the selective SRIs with a neuroleptic or clonazepam.
3. Age between 21 and 65 years.
4. Able to understand and comply with instructions.
5. Able to give fully informed, written consent in the judgment of the site Consent Monitor.
6. Either drug free or on a stable drug regimen for at least 6 weeks.
7. Good general health.
8. A family member or significant other, in contact with the patient every 1-3 days, is available and willing to communicate with the research team if the patient's clinical status worsens, and if necessary to accompany patients to study visits.
9. The local referring psychiatrist is willing to provide ongoing care during and after the trial.
10. Patient is aware of, able to adhere to, and willing to tolerate the frequency of visits associated with adjustment of the dual-stimulation configuration and/or collection of brain recordings. This will usually mean limitation to patients who live close to the study site.
11. Platelet count greater than 125,000 per cubic millimeter and a PT and PTT within normal limits.

Exclusion Criteria:

1. Current or past psychotic disorder.
2. Full-scale IQ below 75 on the Wechsler Abbreviated Scale of Intelligence (WAIS) or cognitive impairment that would affect a participant's ability to give informed consent or provide interview or self-report data reliably, as determined by the consent monitor and the site psychiatrist. A questionnaire assessing consent comprehension will be used with all study subjects, to ensure that they understand the key procedures of the study, and its risks and benefits. An independent monitor will administer that questionnaire.
3. A clinical history of bipolar mood disorder. We will not exclude substance-induced mania or hypomania.

   In our prior studies, a history of induced hypomanic symptoms did not predict DBS-related hypomania.
4. Any current clinically significant neurological disorder or medical illness affecting brain function, other than tic disorders or Tourette syndrome.
5. Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
6. Any labeled DBS contraindication and/or inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia), infection, coagulopathy, inability to undergo an awake operation, significant cardiac or other medical risk factors for surgery.
7. Current or unstably remitted substance abuse, dependence, or a positive urine toxicology screen.
8. Pregnancy and women of childbearing age not using effective contraception.
9. Unable to adhere to operational and administrative study requirements (in the investigators' judgment).
10. Clinical history of severe personality disorder.
11. Imminent risk of suicide or an inability to control suicide attempts (in the investigators' judgment).

    History of serious suicidal behavior or one or more interrupted suicide attempts with potential lethality judged to result in serious injury or death.
12. Diagnosis of body dysmorphic or hoarding disorder.
13. Evidence of dementia or other significant cognitive impairment on neuropsychological evaluation or through cognitive screening (MOCA).

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Yale-Brown Obsessive-Compulsive Scale (YBOCS) | 2 years
  The Yale-Brown Obsessive-Compulsive Scale (YBOCS) will be the principal outcome measure for tracking OCD symptoms. We will collect this measure at all clinical visits.

SECONDARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 2 years
  The Montgomery-Asberg Depression Rating Scale (MADRS) will be a secondary outcome measure for tracking depression symptoms. We will collect this measure at all clinical visits.
Clinical Global Impressions (CGI) Severity and Change scale | 2 years
  The Clinical Global Impressions (CGI) Severity and Change scale will be a secondary outcome measure for tracking global measure of illness severity and change. We will collect this measure at all clinical visits.
Patient Global Impressions (PGI) scale | 2 years
  The Patient Global Impressions (PGI) scale will be a secondary outcome measure for tracking global measure of illness severity and change. We will collect this measure at all clinical visits.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Cusin, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Olsen ST, Basu I, Bilge MT, Kanabar A, Boggess MJ, Rockhill AP, Gosai AK, Hahn E, Peled N, Ennis M, Shiff I, Fairbank-Haynes K, Salvi JD, Cusin C, Deckersbach T, Williams Z, Baker JT, Dougherty DD, Widge AS. Case Report of Dual-Site Neurostimulation and Chronic Recording of Cortico-Striatal Circuitry in a Patient With Treatment Refractory Obsessive Compulsive Disorder. Front Hum Neurosci. 2020 Oct 23;14:569973. doi: 10.3389/fnhum.2020.569973. eCollection 2020. PMID 33192400